CLINICAL TRIAL: NCT03878407
Title: Identification of Patients With Age-Related Clonal Hematopoiesis (ARCH) Among Cancer Survivors.
Acronym: ARCH-001
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: CAPCR 18-5742
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cancer
Keywords: ARCH
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Monitoring of ARCH variants — Blood samples will be tested for mutations, before patients are given Standard of Care chemotherapy/radiation or after given Standard of Care chemotherapy/radiation. Another testing is done after 3 months and after 1 year if positive for ARCH.

SUMMARY:
The purpose of this study is to see if patients with cancer have a certain amount of genetic mutations in their blood. If certain levels of mutations are found in specific genes, patients may have a condition known as ARCH. The prevalence of ARCH is higher in cancer patients who received prior chemotherapy or radiation. Studying ARCH from your blood samples may also help researchers predict which patients are more likely to be prone to heart disease. Patients who are about to start chemotherapy/radiation, and patients who have completed chemotherapy/radiation will be approached to measure the incidence of ARCH. 5-10mL blood samples will be collected before and after treatment, and if ARCH is detected in a laboratory analysis, another blood sample will be collected. Patients with ARCH will repeat the blood collection yearly, and also be referred to a cardiology clinic for follow up.

DETAILED DESCRIPTION:
This is a non-randomized, single-centre, observational study assessing the incidence of ARCH in cancer survivors. Patients over the age of 60 who had or will receive chemotherapy and/or radiation therapy for solid or hematologic malignancies at the Princess Margaret Cancer Centre will be considered. Based on the time point of treatment, patients will either fall into a post or prior chemotherapy/radiation cohort. Peripheral blood will be taken and will be sequenced for ARCH DNA mutations. Patients who have ARCH-related mutations at a variable allele frequency (VAF) of at least 0.5% we will repeat the genetic sequencing yearly to assess changes in mutational spectrum and VAF over time.

ELIGIBILITY:
* Age ≥ 60
* Completed chemotherapy and/or radiation therapy and are being followed at Princess Margaret Cancer Centre i) Patient must be in remission for > 3 months after completing chemotherapy or radiation ii) Predicted 5 year survival of >75% iii) Peripheral blood counts must have returned to normal as defined by:

  1. Platelets ≥ 100 x 109/L
  2. PMN ≥ 1 x 109/L

Or

* Prior to chemotherapy and/or radiation therapy at the Princess Margaret Cancer Centre.
* All histologically/cytologically proven tumour types (solid tumours and hematologic malignancies) will be eligible.
* Received or will receive regimens of chemotherapy or radiation with doses expected to produce transient myelosuppression (PMN<0.5x109/L) in at least 80% of treated patients (The identification and definition of appropriate myelosuppressive chemotherapy and radiation regimens will be at the discretion of the treating physician and will vary among disease sites).
* Patients must have the ability to understand the requirements of the study and provide written informed consent, which includes authorization for release of protected health information
* Patient must be willing to provide a peripheral blood sample.

Exclusion Criteria:

* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 60 who had or will receive chemotherapy and/or radiation therapy for solid or hematologic malignancies at the Princess Margaret Cancer Centre
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Referral to cardiology clinic | 6-12 months

SECONDARY OUTCOMES:
The incidence of ARCH stratified by tumor type. | 6-12 months

OTHER OUTCOMES:
The spectrum of mutations stratified by tumor type. | 6-12 months
The number of patients referred to the ARCH clinic | 6-12 months
The change in VAF over time post chemotherapy/radiation | 6-12 months
The change in VAF pre and post chemotherapy/radiation | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chen, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There's no plan for data sharing outside of the institution.